CLINICAL TRIAL: NCT02611440
Title: Impact of a Pluriprofessional Intervention to Improve Medication Adherence (Secondary Preventive Medication) in Patients After Ischemic Stroke (ADMED-AVC)
Brief Title: Impact of a Pluriprofessional Intervention to Improve Medication Adherence (Secondary Preventive Medication) in Patients After Ischemic Stroke
Acronym: ADMED-AVC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2014.859
Record Dates: First submitted 2015-10-01; First posted 2015-11-20 (Estimated); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Ischemic Stroke
Keywords: ischemic stroke; medication adherence; cardiovascular disease prevention
MeSH Terms: conditions — Ischemic Stroke; Medication Adherence | interventions — Pharmaceutical Services

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pharmacist Intervention (Experimental): It will be a semi -structured interviews with patient and pharmacist over various time after the stroke (at Month0, M3, M6, M9) combined with patient's therapeutic follow-up from various healthcare professionals.
  Interventions: Behavioral: Pharmaceutical care
- Control (No Intervention): No pharmacist intervention planned.

INTERVENTIONS:
Behavioral: Pharmaceutical care — Initial interview with pharmacist (at the hospital discharge): Evaluation aimed to identify barriers to adherence to drug treatment followed by an information session on the disease, the benefit of drugs and the importance of diet and lifestyle habits. Pharmacist advices focused on how to take medication and how to manage adverse events will be provided.
  Telephone interviews with hospital clinical pharmacist - patient (at M3 M6 and M9): The objective is to review with the patient its medication-taking routine and its potential difficulties, to motivate adherence to treatment and lifestyle/dietary rules, to give advices about therapeutics and how to take medication.
  HCP contacts CP to determine the prescription refill. Final interview with HCP pharmacist (at M12): The objective is to take stock with the patient about its taking drug load.
  Arms: Pharmacist Intervention

SUMMARY:
Medication adherence is a major factor to prevent vascular recurrence after a first ischemic stroke. Nevertheless, it is suboptimal and the implementation of specific interventions are needed to improve it.

A patient - centered and pluriprofessional structured intervention, targeting the medication, introduced at hospital discharge and continued at home (by regular telephone contact) could improve medication adherence one year after stroke.

This intervention would consist of semi structured interviews patient-pharmacist at different times during one year after stroke. The information about the therapeutic management of the patient will be shared between healthcare professionals : general practitioners (GP) and community pharmacists (CP), hospital clinical pharmacist (HCP) and physician (HPhys).

It will allow for decrease of the recurrent stroke and others cardiovascular complications based on a better adherence to preventive medication. Furthermore the decrease of the iatrogenic events and the improvement of the quality of life of patients may be also associated.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years
* Patient with ischemic stroke hospitalized in physical medicine and rehabilitation unit or neurovascular unit
* Return at home at the hospital discharge
* Medication including an antiplatelet drug or an oral anticoagulant with at least an antihypertensive drug and/or a lipid lowering agent (statin)
* Patient without either cognitive disorders or major psychiatric disorders
* Patient with a sufficient autonomy for the management of medication at home (score of Barthel > 30)

Exclusion Criteria:

* Patient ≤ 18 years
* Patient with important cognitive or psychiatric disorders
* Management of patient medication exclusively by the helper
* No usual pharmacy (or more than 2 usual pharmacies)
* Patient directed to an institution at the end of the hospitalization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Estimated)
Dates: Start 2015-07-29 (Actual); Primary Completion 2020-07-28 (Estimated); Study Completion 2020-07-28 (Estimated)

PRIMARY OUTCOMES:
Measure of patient's adherence to medication. This adherence measurement is a composite measure | One year after inclusion
  A patient will be considered adherent if:
  1. For each secondary-preventive drug (antiplatelet, lipid lowering, and antihypertensive), evaluated by the pharmacy refills: Number of days of medication available to the patient (supplied by the pharmacy divided by the total number of days in the period of the study (365)), is higher than 80%.
  2. And score obtained from self-reported adherence questionnaire, greater than 6/8 is obtained for all secondary preventative medication

SECONDARY OUTCOMES:
Analysis of pharmacy refills | 1 year after inclusion
  To estimate the benefit of the intervention on the adherence for each drug, number of days of medication available to the patient (supplied by the pharmacy) divided by the total number of days in the period of the study (365) is higher than 80%.
Percentage of patients with drug-related iatrogenic events | 1 year after inclusion
  To estimate the benefit of the intervention on the drug-related iatrogenic events, with a particular attention on the antiplatelet, VKA and the direct oral anticoagulants drugs
Percentage of patients with a new stroke or cardiovascular event | 1 year after inclusion
  To estimate the benefit of the intervention on the recurrence of stroke or another cardiovascular event
Percentage of patients readmitted in hospitalization | 1 year after the inclusion
  To estimate the benefit of the intervention on the rehospitalization
Realization of a questionnaire (Likert-type scale) | 1 year after inclusion
  To estimate the benefit of the intervention on the lifestyle risk factors
Measure of glycemic and lipid balance. | 1 year after inclusion
  To estimate the benefit of the intervention on laboratory tests
Realization of a questionnaire scoring (SF-36 scale) | 1 year after inclusion
  Estimate the benefit of the intervention on the quality of life of the patients
Realization of a questionnaire (Brief IPQR) | 1 year after inclusion
  Estimate the profit of the intervention on the representation of the disease for the patient
Brief IPQR score and medication adherence (treatment adherence score and pharmacy refills) correlation (composite measure) | 1 year after inclusion
  To measure impact of the representation of the disease on adherence to medication
Realization of questionnaires (Likert-type scale and SATMED) assessment of satisfaction of patients | 1 year after inclusion
  To estimate in each groups, the satisfaction of patients on their therapeutic follow-up, on their medication, and their relationship with the healthcare professionals (CP , GP , HCP, HPhys)
Realization of a questionnaire (Likert-type scale) assessment of satisfaction of GP and CP in relation to ADMED-AVC program. | 1 year after inclusion
  To estimate the satisfaction of general practitioners and community pharmacists concerning the ADMED-AVC's program

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - Service de neurologie vasculaire, Hôpital P Wertheimer, HCL, Bron
  - Service de médecine physique et de réadaptation, Hôpital Nord, CHU de Clermont Ferrand, Cébazat
  - Service de médecine physique et de réadaptation, Hôpital sud, CHU de Grenoble, Échirolles
  - Service de médecine physique et de réadaptation, Groupe hospitalier Lariboisière - Fernand Vidal, AP-HP, Paris
  - Service de médecine physique et de réadaptation, Hôpital Bellevue, CHU Saint Etienne, Saint-Etienne
  - Service de médecine physique et de réadaptation, Hôpital Henry Gabrielle, Groupement Hospitalier Sud, HCL, Saint-Genis-Laval

REFERENCES:
- [Derived] Khettar S, Jacquin Courtois S, Luaute J, Decullier E, Bin S, Dupuis M, Derex L, Mechtouff L, Nighoghossian N, Dussart C, Rode G, Janoly-Dumenil A. Multiprofessional intervention to improve adherence to medication in stroke patients: a study protocol for a randomised controlled trial (ADMED AVC study). Eur J Hosp Pharm. 2022 May;29(3):169-175. doi: 10.1136/ejhpharm-2020-002425. Epub 2020 Sep 25. PMID 32978218